CLINICAL TRIAL: NCT03297593
Title: Nivolumab in Combination With Ipilimumab in Patients With Metastatic Renal Cell Carcinoma: A Multicenter Single-arm Phase lI Trial
Brief Title: Nivolumab in Combination With Ipilimumab in Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 07/17
Record Dates: First submitted 2017-09-14; First posted 2017-09-29 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Renal Cell Carcinoma
Keywords: renal cell carcinoma; Nivolumab; Ipilimumab; metastatic renal cell carcinoma; immunotherapy; Opdivo; Yervoy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Prospective single-stage single-arm multicenter phase II trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nivolumab and ipilimumab (Experimental): Patients start treatment with nivolumab (240 mg every 2 weeks during the first 20 weeks, 480 mg every 4 weeks thereafter).
  After 2 weeks, ipilimumab (1mg/kg every 6 weeks) will be introduced. As soon as a radiographic complete response (CR) or partial response (PR) is observed, ipilimumab has to be stopped and only the single-agent treatment with nivolumab is continued. Once ipilumimab has been stopped because of a response, it will not be re-started later on.
  Interventions: Drug: nivolumab; Drug: ipilimumab

INTERVENTIONS:
Drug: nivolumab — 240 mg every 2 weeks during the first 20 weeks, 480 mg every 4 weeks thereafter
  Other Names: Opdivo
Drug: ipilimumab — After 2 weeks 1mg/kg every 6 weeks
  Other Names: Yervoy

SUMMARY:
Immunotherapy with checkpoint inhibitors that target PD-1 and CTLA-4 have shown activity in mRCC. However, the optimal schedule of the combination therapy has yet to be defined.

The objective of the trial is to determine the efficacy of combination immunotherapy of nivolumab and ipilimumab in patients with metastatic renal cell carcinoma.

The expansion phase shall address the role of ipilimumab in case of clinically insignificant progression.

DETAILED DESCRIPTION:
Despite the encouraging results of recent trials, only a minority of patients shows significant response to single agent immunotherapy with nivolumab (Overall response rate (ORR) around 20%). Therefore, further investigations are urgently needed to improve the prognosis of patients with mRCC. Recent analyses of phase I trials in mRCC and also in non-small-cell lung carcinoma (NSCLC) patients as well as more advanced studies in melanoma patients have provided evidence that combination of immunotherapies can improve response rates and response duration.

Cancer immunotherapy rests on the premise that tumors can be recognized as foreign rather than as self and can be effectively attacked by an activated immune system. An effective immune response in this setting is thought to rely on immune surveillance of tumor antigens expressed on cancer cells that ultimately results in an adaptive immune response and cancer cell death. Meanwhile, tumor progression may depend upon acquisition of traits that allow cancer cells to evade immunosurveillance and escape effective innate and adaptive immune responses. Current immunotherapy efforts attempt to break the apparent tolerance of the immune system to tumor cells and antigens by either introducing cancer antigens by therapeutic vaccination or by modulating regulatory checkpoints of the immune system.

Dysfunctional T cells in cancer show an upregulation of inhibitory receptors (T cell exhaustion). Combined blockade of inhibitory receptors including CTLA-4 and PD-1 are considered to act synergistically. Indeed, early trials in mRCC showed improved response rates and combinations have also demonstrated to be prolonging progression-free survival in melanoma. While CTLA-4 is mainly involved in transmitting negative signals in T cells during priming in the lymph node, PD-1 is thought to mainly inhibit T cell cytotoxicity within the tumor by engagement of ligands PD-L1 and PD-L2, which are upregulated by tumor cells and inflammatory cells within the tumor microenvironment as shield against the immune attack. It is therefore reasonable to combine PD-1 blockade with CTLA-4 blockade and this has been tested with an intriguing doubling of ORR in a phase I trial in patients with mRCC. An important aspect of any combination therapy is the question of additional/ excessive toxicity. In that trial the combination of nivolumab 3mg/kg/q3w (cont.) and ipilimumab 1mg/kg/q3w (4 times) proved to be safe, efficacious and feasible (much better safety profile in patients with mRCC compared to patients in melanoma trials). 78% of patients had any AE, but only 28% a grade 3-4 AE event. While diarrhea was quite common, only 4.8% had grade 3-4 diarrhea. Other treatment related immune-mediated AEs, especially endocrinopathy, pneumonitis, skin disorders were recorded at lower grades than 3. No deaths were reported for this combination. The overall response rate was 43% with durable responses of 78% in patients that had an initial response (durable responses).

Moreover, recent variations of dosing schedules and strengths of the nivolumab-ipilimumab combinations have shown improvement of toxicity rates with no loss of efficacy. For example, ipilimumab every 6 weeks at 1mg/kg was shown to be well tolerated in patients with non-small cell lung cancer when combined with nivolumab.

Nivolumab has proven efficacy and a favorable toxicity profile as a 2nd line therapy in mRCC. It is therefore destined to become the standard therapy after a first line TKI therapy. However, only a minority of patients shows clear responses leaving plenty of room for improvement. The addition of a further agent including blockade of CTLA-4 that acts synergistically could improve the response rate and also extend the progression-free and overall survival in patients with mRCC.

The addition of ipilimumab to nivolumab in order to increase response rates and induce more often durable remissions in patients is a reasonable next step and is currently tested in several randomized trials. However, at this point it is unclear which subgroup benefits most from the combination of CTLA-4 and PD-1 blockade and the optimal regimen/schedule remains unknown. To this end, this trial will test a combination of ipilimumab with nivolumab at an alternate schedule and a subsequent adaptation of the treatment regimen to the individual response with the aim to increase efficacy while reducing toxicity in mRCC patients. Ipilimumab is often used only in the first weeks of antineoplastic treatment for initial immune priming, allowing the presumption that it could be stopped after an initial priming phase. A phase I dose finding study is not needed, as experience with this dose and even higher doses have been reported and data are on file at Bristol-Myers Squibb (BMS). In addition, sequential biopsies and biomarker studies shall identify patients that benefit the most of a combination immunotherapy. In this trial, it was decided to have a nivolumab lead-in phase to be able to determine whether any acute side effect is nivolumab or ipilimumab related.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations before registration and prior to any trial specific procedures
* Histologically or cytologically confirmed, locally advanced and/or metastatic clear cell RCC not amenable to surgery or definitive radiotherapy, and requiring systemic therapy
* Patient able and willing to provide serial biopsies and blood drawings (initial, at 14 weeks (except for patient in the expansion cohort), and at progression).
* Measurable disease
* In case of second line patients, the previous therapy must be stopped at least 2 weeks prior to registration
* Age ≥ 18 years
* WHO performance status of 0-1
* Bone marrow function: neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L
* Hepatic function: total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN), AST, ALT and AP ≤ 2.5 x ULN (≤ 5 x ULN if significant hepatic metastasis is suspected to be the cause for enzyme elevation)
* Renal function: eGFR > 20 mL/min/1.732
* Cardiac function: NYHA ≤ 2. In case of cardiac insufficiency NYHA 1 or 2, Left ventricular Ejection Fraction (LVEF) ≥ 35% as determined by echocardiography (ECHO) or multigated acquisition (MUGA) scan
* Women with child-bearing potential are using effective contraception are not pregnant or lactating and agree not to become pregnant during trial treatment and during 5 months thereafter. A negative pregnancy test before inclusion into the trial is required for all women with child-bearing potential.
* Men agree not to father a child during trial treatment and during 5 months thereafter

Exclusion Criteria:

* Uncontrolled CNS metastases. Patients with asymptomatic CNS metastases (at least 2 weeks after radiotherapy or surgery and steroids with prednisone equivalent of 10 mg or lower) are eligible
* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years from registration with the exception of pT1-2 prostate cancer Gleason score < 6, adequately treated cervical carcinoma in situ, or localized non-melanoma skin cancer.
* More than one previous line of systemic therapy for mRCC
* Prior immunotherapy.
* Concurrent or recent (within 30 days of registration) treatment with any other experimental drug
* Concomitant use of other anti-cancer drugs or radiotherapy except for local pain control (radiotherapy of target lesion not allowed)
* Immunosuppressive medications (such as but not limited to: methotrexate, azathioprine, and TNF-α blockers) within 30 days before registration

Exception:

* systemic corticosteroids at doses not exceeding 10 mg/day of prednisone or equivalent
* immunosuppressive medications for patients with contrast allergies
* inhaled and intranasal corticosteroids
* Live attenuated vaccination within 30 days prior to registration and for 30 days after last dose of any of the trial drugs. Inactivated viruses, such as those in the influenza vaccine, are permitted
* History of or active auto-immune disease with the exception of diabetes mellitus type II
* Human immunodeficiency virus (HIV) infection or active chronic Hepatitis C or Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment
* Known hypersensitivity to trial drug(s) or to any component of the trial drug(s)
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | at 2 years.
  ORR is defined as proportion of patients achieving partial response (PR) or complete response (CR) according to RECIST v1.1 at any time between registration and documented disease progression*, death, or subsequent therapy, whichever occurs first.
  *PD before the 3rd administration of ipilimumab not leading to treatment discontinuation does not count as progression for this endpoint. Furthermore, the additional tumor assessment at 20 weeks for patients with PD n.c.s. before week 20 will not be taken into consideration for calculation of this endpoint.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | at weeks 8, 14, 20, 26, and then every 12 weeks up to 2 years.
  PFS is defined as the time from registration until progression according to RECIST v1.1 or death from any cause, whichever occurs first.
  PD before the 3rd administration of ipilimumab not leading to treatment discontinuation does not count as progression for this endpoint. Furthermore, the additional tumor assessment at 20 weeks for patients with PD n.c.s. before week 20 will not be taken into consideration for calculation of this endpoint.
  Patients without event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of the last tumor assessment showing non-progression (before the start of the new therapy, if any).
Duration of response (DOR) | at weeks 8, 14, 20, 26, and then every 12 weeks up to 2 years.
  DOR is defined as time from the date when a patient first meets the criteria for PR or CR according to RECIST v1.1, until documented progression, relapse or death due to disease progression, whichever occurs first.
  PD before the 3rd administration of ipilimumab not leading to treatment discontinuation does not count as progression for this endpoint. Furthermore, the additional tumor assessment at 20 weeks for patients with PD n.c.s. before week 20 will not be taken into consideration for calculation of this endpoint.
  Patients without event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of the last tumor assessment showing non-progression before the start of the new therapy (if any).
  DOR will only be analyzed in the subgroup of patients achieving PR or CR during trial treatment.
Time to treatment failure (TTF) | at weeks 8, 14, 20, 26, and then every 12 weeks up to 2 years.
  TTF defined as time from registration to treatment discontinuation due to any reason. Patients still on treatment at the time of analysis will be censored at the date of last treatment administration. Furthermore, the additional tumor assessment at 20 weeks for patients with PD n.c.s. before week 20 will not be taken into consideration for calculation of this endpoint.
Overall survival (OS) | At weeks 8. 14, 20, 26, then every 12 weeks until 2 years.
  OS is defined as the time from registration until death from any cause. Patients without event at the time of analysis will be censored at the date they were last known to be alive.
Adverse events (AEs) | at weeks 8, 14, 20, 26, then every 12 weeks, until 100 days after last dose of treatment.
  AEs are assessed according to NCI CTCAE v4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Stenner, Prof, Study Chair — Universitätsspital Basel; Heinz Läubli, MD, Study Chair — Universitätsspital Basel
Locations (14):
- Switzerland (14):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Baselland Bruderholz, Bruderholz
  - Kantonsspital Graubünden, Chur
  - Spital Thurgau, Frauenfeld
  - HFR - Hôpital cantonal, Fribourg
  - Hôpitaux Universitaires de Genève, Geneva
  - Centre hospitalier universitaire vaudois - CHUV, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - UniversitätsSpital Zürich, Zurich